CLINICAL TRIAL: NCT06358014
Title: Beijing Anding Hospital Affiliated to Capital Medical University
Brief Title: Assessment of the Improvement in Cognitive Levels of Postmenopausal Depression Patients by Estrogen
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiao Wang (Other)
Responsible Party: Sponsor-Investigator, Xiao Wang, prof, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YX2021-02
Record Dates: First submitted 2024-04-01; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Postmenopausal Depression; Estrogen
MeSH Terms: interventions — Estradiol; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Intervention Model Description: The combination group will receive estrogen combined with Selective serotonin reuptake inhibitors (SSRIs) , while the control group will only receive Selective serotonin reuptake inhibitors (SSRIs) intervention.SSRIs include Citalopram (Celexa) , Escitalopram (Lexapro) ,Fluoxetine (Prozac) ,Paroxetine (Paxil, Pexeva) and Sertraline (Zoloft)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The combination group is estrogen combined with SSRIs for 8 weeks (Experimental): The estradiol/estradiol-norethindrone acetate combination tablet will be taken orally before bedtime, 1 tablet/d (trade name: Fematon, Abbott Laboratories, USA, this product is a combination package, with estradiol 1 mg in the first 14 days of each treatment cycle, and estradiol 1 mg and norethindrone acetate 10 mg in the last 14 days of each treatment cycle). This study uses SSRIs class drugs, including fluoxetine, paroxetine, fluvoxamine, sertraline, citalopram, and escitalopram, with no specific restrictions on the type of drugs.
  Interventions: Drug: Fematon (estradiol/estradiol-norethindrone acetate combination tablet package)+SSRIs
- SSRIs for 8 weeks (Placebo Comparator): This study uses SSRIs class drugs, including fluoxetine, paroxetine, fluvoxamine, sertraline, citalopram, and escitalopram, with no specific restrictions on the type of drugs.
  Interventions: Drug: SSRIs

INTERVENTIONS:
Drug: Fematon (estradiol/estradiol-norethindrone acetate combination tablet package)+SSRIs — In the combination group, eligible subjects will receive 1 tablet/day of estradiol/estradiol-norethindrone acetate combination tablet for 8 weeks. The estradiol/estradiol-norethindrone acetate combination tablet will be taken orally before bedtime, 1 tablet/day (trade name: Fematon, Abbott Laboratories, USA, this product is a combination package, with estradiol 1 mg in the first 14 days of each treatment cycle, and estradiol 1 mg and norethindrone acetate 10 mg in the last 14 days of each treatment cycle). This study uses SSRIs class drugs, including fluoxetine, paroxetine, fluvoxamine, sertraline, citalopram, and escitalopram.
  Arms: The combination group is estrogen combined with SSRIs for 8 weeks
Drug: SSRIs — This study uses SSRIs class drugs, including fluoxetine, paroxetine, fluvoxamine, sertraline, citalopram, and escitalopram, with no specific restrictions on the type of drugs. During the study, medication doses will be quantitatively adjusted based on the results of each visit assessment combined with drug concentrations.
  Arms: SSRIs for 8 weeks

SUMMARY:
After menopause, there is a certain tendency towards depression, with the risk of developing depression being about 3 to 4 times higher than before menopause. Additionally, postmenopausal women experience varying degrees of cognitive decline, which are closely associated with hormonal changes. Therefore, we should pay more attention to the cognitive levels of postmenopausal depression patients. Increasing evidence suggests that changes in cognitive function during menopause may be related to the effects of estrogen on cognitive function, and estrogen therapy can effectively improve cognitive decline. Estrogen is not only associated with cognitive symptoms after menopause, but estrogen intervention is also an adjunctive treatment for postmenopausal depression symptoms. There is a close relationship between cognitive levels and depression, as depression itself is accompanied by cognitive decline, and early cognitive decline can also manifest depressive symptoms. Therefore, the cognitive levels of postmenopausal depression patients are also worthy of further attention.This study is an 8-week randomized controlled trial. The subjects are patients with postmenopausal depression accompanied by cognitive decline, all of whom have undergone natural menopause for at least one year; with HAMD-17 scores ≥17 points; and MOCA scores ≤26 points. This study aims to recruit patients with postmenopausal depression accompanied by cognitive decline from the outpatient or inpatient departments of Beijing Anding Hospital, Capital Medical University. Patients who meet the inclusion criteria will be randomly assigned to the combination group and the control group using a random number method. The combination group will receive estrogen combined with SSRIs, while the control group will only receive Selective serotonin reuptake inhibitors (SSRIs) intervention. Patients' cognitive function and depressive symptoms will be assessed using scales at baseline, 2 weeks, 4 weeks, and the end of 8 weeks of treatment, and safety evaluations will be conducted. The primary efficacy endpoint is the change in MoCA scores from baseline to the end of the study. Secondary efficacy endpoints include changes in HAMD-17, modified Kupperman Scale, ADL Scale, and hormone levels from baseline to the end of the study. The safety of the study drug will be evaluated through adverse event reporting, clinical laboratory tests, and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients from outpatient or inpatient departments;
2. Patients who sign a written informed consent form;
3. Natural menopause for at least 1 year, with first-onset depression, aged ≤70 years;
4. Meeting the diagnostic criteria for Major Depressive Disorder according to the Diagnostic and Statistical Manual of Mental Disorders-fifth Edition (DSM-5);
5. HAMD-17 score ≥17 points;
6. Presence of cognitive impairment symptoms, Montreal Cognitive Assessment scale (MoCA) <26 points;
7. Education level of primary school or above.

Exclusion Criteria:

1. Patients with significant physical illness, cranial trauma, or other serious unstable physical illnesses;
2. Patients who have participated in another interventional clinical study in the past month;
3. History or current diagnosis of the following psychiatric disorders according to DSM-5: organic mental disorders, Alzheimer's disease, other causes of secondary dementia, schizophrenia, schizoaffective disorder, bipolar affective disorder, delusional disorder, unspecified mental disorders, patients with a history of substance abuse, including alcohol and active substance abuse in the past 12 months, excluding nicotine;
4. Currently taking antidepressants, cognitive enhancers, or other psychiatric medications in the past 2 weeks;
5. Severe speech, visual, or hearing impairments that prevent completion of scale assessments;
6. Individuals with severe suicidal ideation or suicidal behavior;
7. Patients with malignant tumors;
8. Known or suspected history of breast cancer;
9. Known or suspected estrogen-dependent malignant tumors (such as endometrial cancer);
10. Known or suspected progesterone-dependent tumors;
11. Untreated endometrial hyperplasia;
12. Unexplained vaginal bleeding.

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The average change value of MOCA total scores from baseline to 8 weeks of treatment, as assessed by raters, is the primary efficacy endpoint(0-8week). | 8 week
  Montreal Cognitive Assessment (MoCA) Test is based on scores with a maximum score of 30. It takes 10 to 12 minutes to complete.The cutoff for a normal MoCA score is 26. Scores of 25 and below may indicate mild cognitive impairment.

SECONDARY OUTCOMES:
The average change value of HAMD-17 total scores from baseline to 8 weeks of treatment, as assessed by raters, is secondary Outcome Measures | 8 week
  Hamilton Depression Rating Scale (HAMD-17) is scored by summing the item scores. The total score can range from 0 to 54, with higher scores indicating a greater severity of depression. 0 - 7 = Normal. 8 - 13 = Mild Depression. 14-18 = Moderate Depression. 19 - 22 = Severe Depression. > 23 = Very Severe Depression
The average change value of HAMA total scores from baseline to 8 weeks of treatment, as assessed by raters, is secondary Outcome Measures | 8 week
  Hamilton Anxiety Rating Scale (HAMA) ,Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indi- cates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
The average change value of Kupperman total scores from baseline to 8 weeks of treatment, as assessed by raters, is secondary Outcome Measures | 8 week
  The Blatt-Kupperman menopausal index included 11 symptoms which were rated on a four point scale from 0=none to 3=severe. These ratings were then summed across the 11 items and the score was categorized as follows: none 0-5, mild 5-10, moderate 10-15, severe 15+.
The average change value of PSQI total scores from baseline to 8 weeks of treatment, as assessed by raters, is secondary Outcome Measures | 8 week
  Pittsburgh Sleep Quality Index (PSQI) Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
The average change value of ADL total scores from baseline to 8 weeks of treatment, as assessed by raters, is secondary Outcome Measures | 8 week
  Activities of Daily Living (ADL) scores of 0-20 indicate "total" dependency scores of 21-60 indicate "severe" dependency scores of 61-90 indicate "moderate" dependency scores of 91-99 indicate "slight" dependency most studies use a score of 60/61 (moderate dependency) as a cutting point

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anding Hospital Affiliated to Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No
"We currently have no plans to provide Individual Participant Data (IPD) to other researchers."